CLINICAL TRIAL: NCT05009381
Title: A No-treatment Controlled, Prospective, Randomized, Multimulti-center, Evaluator-Blinded Study to Evaluate the Effectiveness and Safety of STYLAGE® XXL for Chin Augmentation in Chinese Adults
Brief Title: Effectiveness and Safety of STYLAGE® XXL for Chin Augmentation in Chinese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Vivacy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VIV-STYL-XXL-01
Record Dates: First submitted 2021-07-16; First posted 2021-08-17 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Esthetic
Keywords: Chin; Hyaluronic Acid; volume; HA fillers

STUDY DESIGN:
Intervention Model Description: A no-treatment Controlled, Prospective, Randomized, Multimulti-center, Evaluator-Blinded Study
Who Masked: Outcomes Assessor
Masking Description: The primary hypothesis of this trial will be based on the chin volume change assessed by a central reader blinded to subject treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Treatment group will receive STYLAGE® XXL at enrollment with an optional touch up injection 30 days later
  Interventions: Device: Stylage XXL at enrollment
- control group (Experimental): Control group will not be treated at enrollment visit. Subjects will receive STYLAGE® XXL at visit 6 months after randomization, if they are still eligible for chin augmentation with an optional touch up injection 30 days later.
  Interventions: Device: Stylage XXL at Month 6

INTERVENTIONS:
Device: Stylage XXL at enrollment — Injection in the chin at enrollment
  Arms: Treatment group
Device: Stylage XXL at Month 6 — Injection in the chin 6 months after randomization
  Arms: control group

SUMMARY:
The aim of this trial is to demonstrate the efficacy and safety of STYLAGE® XXL in augmenting the chin volume among Chinese adults.

Subjects will be randomized either to the treatment group or the control group in a 4:1 ratio

The superiority of STYLAGE® XXL against no-treatment control in chin volume augmentation will be verified together with assessments of the safety profiles.

DETAILED DESCRIPTION:
This study is a no-treatment controlled, prospective, randomized, multi-center, evaluator-blinded study, in Chinese subjects seeking for chin volume augmentation.

150 subjects will be randomized either to the treatment group or the control group in a 4:1 ratio (120 subjects in the treatment group and 30 subjects in the control group).

Subjets assigned to the treatment group will receive STYLAGE® XXL at enrollment.

Subjects assigned to the control group will not receive treatment at enrollment; however, at 6 month visit, subjects who are still eligible for chin augmentation with STYLAGE® XXL will be treated

STYLAGE® XXL superiority will be demonstrated against no-treatment control in augmenting the chin volume, as measured by blinded evaluator at 6-month

ELIGIBILITY:
Inclusion Criteria:

* Chinese ethnicity
* Subjects seeking for chin volume augmentation
* Per Investigator's assessment, subjects who require 1 to 4 mL total volume of STYLAGE® XXL for chin augmentation to achieve a meaningful improvement and/or change in their aesthetic appearance.
* With realistic expectations who can understand and comply with the instructions and all visit schedule.
* Willing to abstain from other facial cosmetic procedures (e.g., further augmentation therapy, botulinum toxin injections, laser or chemical skin resurfacing, or face lift procedures) below the level of the horizontal line from subnasale for the duration of the study.
* Women of childbearing potential (WOCBP) who agree contraception during the study period.
* Subjects who voluntarily decided the participation of the study and signed the informed consent.
* Being able to stand mild pain.

Exclusion Criteria:

* Subjects who are contraindicated to injection with HA fillers.
* Subjects who had a history of keloid formation or hypertrophic scar.
* Subjects presenting a scar or skin disorder (e.g., active dermal disease [facial psoriasis, eczema, rosacea, perioral dermatitis, acne, herpes, etc], inflammation or an unhealed wound) below the level of the horizontal line from subnasale that may confound the study evaluation.
* Has ever received permanent (non-biodegradable) or semi-permanent fillers or permanent facial implants (e.g., calcium hydroxyapatite, poly-L-lactic acid, polymethylmethacrylate, silicone, expanded polytetrafluoroethylene), or fat injections below the level of the horizontal line from subnasale, or is planning to be implanted with any of these products at any time during the study.
* Has undergone temporary dermal filler treatment (e.g., hyaluronic acid or collagen) for facial tissue augmentation therapy in the chin and/or lips within 12 months before enrollment or is planning to undergo such treatment during the study
* Has undergone botulinum toxin injections, mesotherapy, or cosmetic facial procedures (e.g., facial liposuction, aesthetic surgery, face-lift, photomodulation, intense pulsed light, radio frequency, dermabrasion, laser or chemical peel, or other ablative procedures) below the level of the horizontal line from subnasale within 6 months or is planning to undergo any such treatment during the study.
* Subjects who has any history of severe multiple allergies or an allergy resulting in anaphylaxis, or a hypersensivity to hyaluronic acid and/or one of the ingredients of the study products.
* Subject is pregnant or planning to be pregnant during the study period or lactating. Women of childbearing potential who have a positive pregnancy test result during screening or at baseline. Women of childbearing potential who are unwilling to use effective birth control measures during the full course of the study.
* Subject currently suffering from a serious or progressive disease, which, in the investigator's judgment, put the subject at undue risk for participation in this clinical trial (e.g., cancer or pre-cancer, uncontrolled diabetes, epilepsy, severe cardio-cerebrovascular disease(s) (e.g., stroke, idiopathic aortic stenosis, aneurysm, hypertrophic obstructive cardiomyopathy, ischaemic heart disease, tachyarrhythmias, severe heart failure [classified as NYHA III-IV], etc.) etc.).
* Subjects having history of cancer within 5 years
* Subjects who received oral surgery (e.g., tooth extraction, orthodontia or implantation) or sinus surgery within 6 weeks before enrollment or is planning to undergo any of these procedures during the study.
* Subject has history or active autoimmune disease (e.g., inflammatory bowel disease), active or history of connective tissue disease (rheumatoid arthritis, scleroderma, and systemic lupus erythematosus)
* Subjects with current or a history of hemorrhagic diseases.
* Subjects who received chemotherapy, immunosuppressive agents, immunomodulatory therapy (e.g., monoclonal antibodies), systemic corticosteroids within 3 months before treatment (inhaled corticoids are allowed).
* Subjects unlikely to achieve a meaningful aesthetic result with the prescribed dosage regimen of the study product per Investigator's judgement.
* Subjects who participated in other clinical trial within 30 days or who is in an exclusion period of one (e.g., in the screening period of another trial).
* Subjects with hypertension (systolic blood pressure above 160mmHg or diastolic blood pressure above 100 mmHg at resting status), and/or significant liver (serum ALT or AST ≥2X the upper limit of the reference range), kidney (BUN, Urea or Cr≥1.5X the upper limit of the reference range), and/or blood coagulation disorders (PT, APTT or INR >20% of the reference range).
* Current or a history of alcoholism, drug abuse, or drug dependence
* Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship.
* Subject with a past history of streptococcal disease (manifested by recurrent sore throat or acute rheumatic fever) or with an active infection to streptococcus.
* Has facial hair (e.g., beards, sideburns, etc.), piercing or tattoo in the area to be treated that would interfere with investigation assessments and create inconsistency in required investigation photography during the study period
* Personnel of the study department, close relatives of the study site personnel (e.g., parents, children, siblings, or spouse), employees, or close relatives of employees at the Sponsor or CRO company.
* Other conditions the Investigator considers inappropriate for enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Chin volume change in ml | 6 months
  Chin volume change in ml, from baseline to 6 months (after last treatment in the treatment group, and after randomization in the control group) between the treatment and control groups as measured by the blinded evaluator using the 3D system.

SECONDARY OUTCOMES:
Chin volume change in ml | 3 months
  Chin volume change in ml, from baseline to 1- and 3- months (after last treatment in the treatment group, and after randomization in the control group), respectively, between the treatment and control groups as measured by the blinded evaluator using the 3D system
Glabella-subnasale-pogonion angle change in degrees | 1,3 and 6 months
  Glabella-subnasale-pogonion angle change in degrees, from baseline to 1-, 3-, and 6- months (after last treatment in the treatment group, and after randomization in the control group), respectively, between the treatment and control groups as measured by the blinded evaluator using the 3D system
Global Aesthetic Improvement Scale (GAIS) Optimal chin augmentation defined as the best possible aesthetic result assessed by the Treating investigator | 1,3 and 6 months
  Percentage of responders, defined by having "Improved", "Much improved" or "Very much improved" according to the Treating Investigator assessed Global Aesthetic Improvement Scale (GAIS), at 1-, 3-, and 6- months (after last treatment in the treatment group, and after randomization in the control group), respectively, between the treatment and control groups.
Global Aesthetic Improvement Scale (GAIS) Optimal chin augmentation defined as the best possible aesthetic result assessed by the subject | 1,3 and 6 months
  Percentage of responders, defined by having "Improved", "Much improved" or "Very much improved" according to the Subject assessed Global Aesthetic Improvement Scale (GAIS), at 1-, 3-, and 6- months (after last treatment in the treatment group, and after randomization in the control group), respectively , between the treatment and control groups.
Subject satisfaction assessment | 1,3 , 6 , 9 , 12 months
  Percentage of satisfied subjects on each question of the subject satisfaction questionnaire The response scale for each question consists of five categories (strongly agree, agree, not sure, disagree, strongly disagree). A subject will be considered as "satisfied" if the answer is "strongly agree" or "agree" in that question.
Results of device performance evaluation respectively. | Day 1 and 1 month
  The Treating Investigator will be asked to rate the: (1) ease of injection, (2) extrusion force, and (3) moldability/malleability on an 11-point numeric scale ranged from 0 (Easy) to 10 (Hard)
Safety : report of AE / SAEs | 1,3,6 months
  Adverse Events (AEs) report throughout the study
Safety : Vital signs Body temperature | Screening, Day 1, 1,3,6,9,12 months
  Body temperature will be measured and recorded in degrees Celsius
Safety : Vital signs Heart rate | Screening, Day 1, 1,3,6,9,12 months
  Heart rate : Subjects should be seated at rest to measure heart rate . Heart rate measurements should be made by counting heartbeats for a period of 30 seconds and multiplying these values by 2 to obtain the rates per minute
Safety : Vital signs respiration rate | Screening, Day 1, 1,3,6,9,12 months
  Respiration rate :Subjects should be seated at rest to measure respiratory rate.. Respiration rate will be recorded by counting the number of breath cycles in 1 minute.
Safety : Vital signs Blood pressure | Screening, Day 1, 1,3,6,9,12 months
  Blood pressure (systolic and diastolic) : Blood pressure will be measured in sitting position at rest using a standardized sphygmomanometer equipped in the site and standardized cuff adapted to the size of the subject's arm. The blood pressure is recorded in millimeters of mercury (mmHg)
Safety : Physical evaluation | screening and 12 months
  The physical evaluation is a test to determine the overall health of the subject. The investigator will inspect the following parts of body : Skin and mucous, lymph nodes, head (eyes, nose, ears, mouth), neck (thyroid, vessels, trachea) , chest (heart, lungs), abdomen (liver, spleen, kidney) , muscle-skeleton and neurologic systems by checking consistency,location, size, tenderness, and texure of the individual organs.
Safety : Physical evaluation BMI | screening and 12 months
  Height is measured in meter, weight is measured in kg, BMI is calculated in kg/m^2 where kg is a person's weight in kilograms and m2 is their height in metres squared.
Safety : Physical evaluation Visual inspection of the skin | 1 month
  Visual inspection of the skin in the injection area (e.g., sclerosis, pruritus, pain, reddish, edema, bruises, ecchymosis, infection, inflammation, allergy, and formation of scar and/or granuloma, etc.).
Safety : Clinical Laboratory evaluation PT and APTT | Screening, 1 month , 12 months
  Blood coagulation: PT(prothrombin time), and APTT (activated partial thromboplastin time) are measured in seconds
  Urinalysis: pH, leucocytes, nitrites, protein, blood, glucose Pregnancy testing
Safety : Clinical Laboratory evaluation INR | Screening, 1 month , 12 months
  INR (international normalized ratio) is calculated as a ratio of the patient's PT in seconds to a control PT standardized in seconds
Safety : Clinical Laboratory evaluation FIB | Screening, 1 month , 12 months
  FIB (Fibrinogene) is measured in g/L
Safety : Clinical Laboratory evaluation Glucose and electrolytes | Screening, 1 month , 12 months
  Blood Glucose and serum electrolytes (Na+、K+、Cl-、Ca2+, Mg2+) are measured in mmol/L
Safety : Clinical Laboratory evaluation Hepatic function | Screening, 1 month , 12 months
  ALT/AST aminotransferase enzymes are measured in units/L of serum
Safety : Clinical Laboratory evaluation Renal function | Screening, 1 month , 12 months
  BUN (blood urea nitrogen) and plasma creatinine in mg/dL
Safety : Clinical Laboratory evaluation Hematology cells | Screening, 1 month , 12 months
  RBC count, WBC count with differential are expressed in cells/ mcL (including absolute WBC count, absolute count and percentage of the 5 WBC differentials including neutrophil, eosinophil, basophil, lymphocyte, and monocyte)
Safety : Clinical Laboratory evaluation hematology Hb | Screening, 1 month , 12 months
  Hb (hemoglobin) in g/dL
Safety : Clinical Laboratory evaluation hematology HCT | Screening, 1 month , 12 months
  HCT (hematocrit) in %
Safety : Clinical Laboratory evaluation Hematology PLT | Screening, 1 month , 12 months
  PLT count (platelets/mcL)
Safety : Clinical Laboratory evaluation Urinalysis pH | Screening, 1 month , 12 months
  pH
Safety : Clinical Laboratory evaluation Urinalysis leucocytes | Screening, 1 month , 12 months
  leucocytes in wbc/hpf.
Safety : Clinical Laboratory evaluation Chemical Urinalysis | Screening, 1 month , 12 months
  nitrites, protein, blood, glucose : dispstick urinalysis
Safety : Clinical Laboratory evaluation Pregnancy testing | Screening, 1 month , 12 months
  β-hCG in urine or serum (mIU/mL)
Safety : ECG | Screening, 1 month
  Standard ECGs (12-Lead ECG or 15 Lead ECG) will be recorded in a supine position at resting status

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wu, Principal Investigator — Peking University First Hospital
Locations (5):
- China (5):
  - Beijing Hospital, Beijing, Dong Cheng District
  - Guangdong Second Provincial General Hospital, Guangzhou, Guangdong
  - Peking University Third Hospital, Beijing, Haidian District
  - West China Hospital of Stomatology Sichuan University, Chengdu, Sichuan
  - Peking University First Hospital, Beijing, Xicheng District